CLINICAL TRIAL: NCT03584607
Title: Insulin- and Glucose Metabolism in Pulmonary Arterial Hypertension - a Pilot Study
Brief Title: Insulin- and Glucose Metabolism in Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-066 ex 16/17
Record Dates: First submitted 2018-05-14; First posted 2018-07-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Pulmonary Arterial Hypertension patients: Blood sampling Insulin resistance-measurement
- Healthy controls: Blood sampling Insulin resistance-measurement

SUMMARY:
Insulin resistance is a key mechanism in metabolic disorders, which has also been implicated in the development of pulmonary hypertension. In this pilot study, the investigators´ goal is to directly determine insulin sensitivity in idiopathic pulmonary arterial hypertension patients and to compare the results with data from healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form
* patients with idiopathic or hereditary pulmonary hypertension / healthy controls

Exclusion Criteria:

* premenopausal women
* other relevant lung disease
* relevant left heart disease
* untreated systemic hypertension
* Diabetes mellitus
* pulmonary hypertension other than idiopathic or hereditary form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls, or patients with idiopathic or hereditary pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 1 day
  Determination of insulin sensitivity using hyperinsulinemic-euglycemic clamp technique

CONTACTS AND LOCATIONS:
Overall Officials: Bence M. Nagy, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria

REFERENCES:
- [Derived] Nagy BM, Kovacs G, Tornyos A, Svehlikova E, Foris V, Nagaraj C, Kwapiszewska G, Pieber TR, Olschewski A, Olschewski H. No indication of insulin resistance in idiopathic pulmonary arterial hypertension with preserved physical activity. Eur Respir J. 2020 Jun 11;55(6):1901228. doi: 10.1183/13993003.01228-2019. Print 2020 Jun. No abstract available. PMID 32217652